CLINICAL TRIAL: NCT05999656
Title: Clinical Study on the Safety and Efficacy of Local Injection of Human Cord Blood Mononuclear Cells in the Treatment of Refractory Diabetic Foot
Brief Title: Human Cord Blood Mononuclear Cells in the Treatment of Refractory Diabetic Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Shandong Qilu Stem Cells Engineering Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-752
Record Dates: First submitted 2023-06-27; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Refractory Diabetic Foot; Human Cord Blood-derived Mononuclear Cells; Efficacy; Safety; Local Injection
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- human cord blood-derived mononuclear cells (HCB-MNCs) (Experimental): About 1×10^8 of HCB-MNCs were injected 3 times at a week interval for each participant.
  Interventions: Biological: human cord blood-derived mononuclear cells (HCB-MNCs)

INTERVENTIONS:
Biological: human cord blood-derived mononuclear cells (HCB-MNCs) — All patients received cell therapy for the first time. HCB-MNCs were injected subcutaneously or intramuscularly into the ulcers of the patients' feet, with an interval of about a centimeter between every two points and an injection volume of 0.2ml at each puncture point. The total injection volume required by the patients was the injection needles multiply 0.2ml (about 2ml of suspended cell in total). The remaining suspension was injected on both sides of the center of the main ischemic site. All patients received three injections of umbilical cord blood mononuclear cells at a week interval, with the latter two injections located around the site of the first injection. The adjuvant therapy remained unchanged within two weeks after cell injection. The follow-up period is 12 weeks after treatment to observe safety and efficacy. If the patient does not recover after 12 weeks, the follow-up period can be extended to 24 weeks.

SUMMARY:
Refractory diabetic foot is one of the most serious and costly chronic complications of diabetes. It is the leading cause of nontraumatic lower-extremity amputations while the conventional treatment is not effective. Therefore, new therapeutic methods are urgently needed. Cell therapy has shown unique advantages and potential in tissue regeneration and wound repair, and is considered as a new effective method to treat diabetic foot. Meanwhile, human cord blood-derived mononuclear cells (HCB-MNCs) with its sufficient sources, strong ability of proliferation and differentiation, and weak immunogenicity, is suitable for the treatment of diabetic foot. It is a prospective, single-arm, single-center clinical study to investigate the efficacy and safety of local injection of HCB-MNCs in the treatment of refractory diabetic foot.

DETAILED DESCRIPTION:
Refractory diabetic foot is one of the most serious and costly chronic complications of diabetes, and is the leading cause of nontraumatic lower-extremity amputations. Conventional treatment is symptomatic supportive treatment such as controlling blood sugar, fighting infection, improving blood circulation, using topical medications, etc. But the effectiveness is barely satisfactory, while the wound heals slowly, and the large blood vessels that have been blocked cannot be re-opened. Therefore, an effective method is needed to relieve lower limb ischemia, promote ulcer healing and shorten the treatment time.

Cell therapy has shown unique advantages and potential in tissue regeneration and wound repair, and is considered as a new effective method to treat diabetic foot. Cell treatment for diabetic foot include local injection, intravenous infusion and arterial infusion. At present, local intramuscular injection is used in most studies at home and abroad.

HCB-MNCs is composed of immature immune cells and pluripotent stem cells, which is adequate, superior proliferative and immature , is a favorable source of cells for the treatment of diabetic foot. A few clinical studies have found that local intramuscular injection of HCB-MNCs or combined with gel dressing can effectively treat diabetic foot ulcers and relieve pain and other symptoms of patients. In this study, 24 patients with refractory diabetic foot will be enrolled. HCB-MNCs will be injected into the diabetic foot wound area 3 times at a week interval to explore its effectiveness and safety.

The primary objective of this study is to investigate the safety of local application of HCB-MNCs in the treatment of refractory diabetic foot and the change of wound area. The secondary objective is to assess changes in the visual analogue scale, total symptoms score and wagner scale.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-80 years;
2. Meet the diagnostic criteria of diabetic foot by International Clinical Guidelines for Diabetic Foot;
3. Ulcer course ≥8 weeks, Wagner grade ≥2;
4. There was no healing trend (no reduction in wound size and no obvious new granulation tissue) after 4 weeks or above treatment. Or the ulcer was further aggravated (by Wagner's grade assessment) in the course of standardized treatment;
5. Fasting blood glucose ≤9mmol/L, 2h postprandial blood glucose ≤13mmol/L;
6. Signing informed consent.

Exclusion Criteria:

1. Patients with a history of ketoacidosis and hyperosmosis within 6 months;
2. Patients with viral infection (treponema pallidum, active hepatitis, HIV, Epstein-Barr virus, etc.)
3. Patients with malignant disease or cured of basal cell carcinoma within the past 5 years;
4. Creatinine clearance < 45ml/min;
5. Patients with severe heart failure (NYHA III-IV);
6. Patients with a history of myocardial infarction or cerebral infarction in the last 3 months;
7. Patients who have received cell or growth factor therapy in the past year;
8. Patients during pregnancy or lactation;
9. Patients with abnormal thyroid dysfunction history or abnormal control through drug treatment;
10. Patients with severe hepatic failure (ALT, AST: above 3 times the upper limit of normal);
11. Lower extremity arterial with large artery occlusion by ultrasound image;
12. Patients with a history of severe coagulation disorder or hemorrhagic disease;
13. Patients with sequelae of cerebral infarction or other reasons that cannot extend their lower limbs flat;
14. Patients with psychological or mental disorders who cannot cooperate with treatment;
15. Participate in other clinical research within the past three months;
16. Patients are unable to complete the study or comply with the requirements of the study by investigator's judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05-28 (Actual); Primary Completion 2024-05-28 (Estimated); Study Completion 2024-11-28 (Estimated)

PRIMARY OUTCOMES:
Number of patients with no adverse reactions. | From baseline to 12 weeks after the first treatment. The follow-up period can be extended up to 24 weeks if the patient's foot ulcers have not healed at 12 weeks.
  The patient completed 3 times HCB-MNCs treatment and follow-up, and there were no adverse reactions that needed to be stopped. Adverse reactions refer to any symptoms, syndromes or diseases that affect patients' health during clinical research and observation, and also include clinically relevant situations found in the laboratory or other diagnostic processes, such as unplanned diagnosis and treatment measures, withdrawal from research, or clinically significant laboratory examination items. Blood routine, fasting blood glucose, postprandial blood glucose, blood biochemistry, coagulation function, tumor markers and adverse reactions will be recorded during the follow-up.
Rate of wound area change | From baseline to 12 weeks after the first treatment. The follow-up period can be extended up to 24 weeks if the patient's foot ulcers have not healed at 12 weeks.
  The changes of ulcer wound area were compared weekly before and after local application of HCB-MNCs until the wound heals or the follow-up period ends or the wound area no longer changes. The formula for calculating the change rate of periwound is:
  Rate of wound area change=(Wound area per week after treatment-Area of wound before treatment)/ Area of wound before treatment×100

SECONDARY OUTCOMES:
Change in visual analogue scale (VAS) | From baseline to 12 weeks after the first treatment. The follow-up period can be extended up to 24 weeks if the patient's foot ulcers have not healed at 12 weeks.
  A Recognized scale containing scores from 0 to 10, with higher scores indicating a worse outcome.
Change in total symptoms score (TSS) | From baseline to 12 weeks after the first treatment. The follow-up period can be extended up to 24 weeks if the patient's foot ulcers have not healed at 12 weeks.
  A Recognized scale containing scores from 0 to 4, with higher scores indicating a worse outcome.
Change in Wagner scale | From baseline to 12 weeks after the first treatment. The follow-up period can be extended up to 24 weeks if the patient's foot ulcers have not healed at 12 weeks.
  A Recognized scale containing levels from 0 to 5, with higher levels indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Yang, Study Chair — The First Affiliated Hospital with Nanjing Medical University; Xuqin Zheng, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No
The medical records of the subjects (research medical records , laboratory sheets, etc.) will be kept intact in the hospital. The project researchers, ethics committee and project funding department will be allowed to consult the medical records of the subjects. Any public report on the results of this study will not disclose the personal identity of the subjects. We will make every effort to protect the privacy of the subjects' personal medical data within the scope permitted by the laws of the People's Republic of China.